CLINICAL TRIAL: NCT05938218
Title: Virtual Reality Assisted Patient Empowerment: Diagnose ATTR-Amyloidosis And Start Treatment
Acronym: VRAP-DAAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Record Dates: First submitted 2023-06-20; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Amyloidosis Cardiac; Virtual Reality
Keywords: ATTR; cardiac amyloidosis; Virtual Reality; Suspected transthyretin amyloid cardiomyopathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Methods

STUDY DESIGN:
Intervention Model Description: In this intervention, VR glasses with an information module are utilized, lasting approximately 25 minutes. This intervention takes place in the waiting room prior to the actual physician-patient conversation and complements the usual care provided through brochures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): In this intervention, VR glasses with an information module are utilized, lasting approximately 25 minutes. This intervention takes place in the waiting room prior to the actual physician-patient conversation and complements the usual care provided through brochures
  Interventions: Device: Intervention
- Control Group (No Intervention): Usual Care

INTERVENTIONS:
Device: Intervention — Virtual Reality assisted information Patients in the intervention group receive a VR instructional application lasting approximately 25 minutes. This intervention takes place in the waiting room prior to the actual physician-patient conversation and complements the usual care provided through brochures.
  Arms: intervention

SUMMARY:
ATTR amyloidosis is a serious condition with significant morbidity and mortality. In Germany, there are numerous unreported cases of untreated patients, and diagnosing and initiating treatment often requires multiple specialized tests. To address this, a study is being conducted to determine if virtual reality (VR)-based patient education can improve diagnosis rates, treatment initiation, and medication adherence compared to standard education methods.

DETAILED DESCRIPTION:
Tafamidis is effective in reducing mortality and hospitalization in patients with transthyretin amyloid cardiomyopathy (ATTR-CM), and adherence to the drug is generally high. However, the main challenge lies in timely diagnosis and initiation of therapy. Virtual reality (VR) offers an immersive educational tool that surpasses conventional methods like brochures and videos, with patients preferring VR glasses. By preparing patients through VR, they can engage in informed conversations with physicians, understand the diagnostic process better, and be motivated to initiate therapy promptly. VR empowers patients and saves valuable time for physicians, and it has been well-received even among older cardiovascular patients

ELIGIBILITY:
Inclusion Criteria:

* patients who present themselves for assessment of an unclear septal thickening with suspicion of cardiac amyloidosis.

Exclusion Criteria:

1. < 18 years
2. Active Medication with tafamidis
3. Cardiovascular Disease
4. highly impaired vision or hearing
5. advanced dementia syndrome
6. epilepsy
7. insufficient language skills

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time-to-Event | up to 180 days
  Count days after first use of VR until the final diagnosis or prescription of tafamidis is given. [time frame: xx days]
  1. Time-to-Event [days] Count days after first use of VR until the final diagnosis or prescription of tafamidis is given. [time frame: xx days]
  Count days after first use of VR until the final diagnosis or prescription of tafamidis is given

SECONDARY OUTCOMES:
Duration patient-physician talk | up to 30 minutes
  Duration of the patient-physician talk in minutes.
Drug-Adherence to tafamidis | after 6 months after enrollment
  Drug-Adherence to tafamidis (yes/no/unknown)
health literacy: Baseline | 1 hour before patient-physician talk after enrollment
  In order to test to assess the health literacy at baseline, a health literacy questionnaire will be asked
Health literacy: after the first patient-physician-talk | 1 hour after patient-physician talk]
  In order to test to what extent the addition of a combination of different learning modalities (acoustic, visual, written, haptic) implemented in virtual reality to the medico-legal informed consent is superior to the standard informed consent, a survey is conducted after the informed consent using a health literacy questionnaire
Health literacy baseline: Long term | up to 180 days after patient-physician talk
  In order to test to what extent the addition of a combination of different learning modalities (acoustic, visual, written, haptic) implemented in virtual reality to the medico-legal informed consent is superior to the standard informed consent, a survey is conducted after the informed consent in terms of long term effects using a health literacy questionnaire
Rate of patients who died or were re-hospitalized during the long term follow up | after 6 and 12 months after enrollment
  patients are contacted and information is gathered about survival of the patients and possible rehospitalization events due to cardiac events
Kansas City Cardiomyopathy Questionnaire (KCCQ) | after 6 months after enrollment
  KCCQ will be used to assess the general the patient's perception of their health status. In the KCCQ-12, responses are given on a Likert scale that for each individual item is scored on a scale of 0-100 with higher scores indicating better health
Simulator Sickness Questionnaire (SSQ) | immediately after Virtual Reality (VR-) Education
  A SSQ will assess for VR associated compatibility. SSQ asks participants to provide subjective severity ratings of 16 symptoms on a scale from 0 (no perception) to 3 (severe perception) after the exposure. Total scores can be associated with negligible (< 5), minimal (5 - 10), significant (10 - 15), and concerning (15 - 20) symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jung, Prof. Dr., Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- University-Hospital Düsseldorf Division of Cardiology, Pulmonary Disease and Vascular Medicine [Recruiting] Düsseldorf, Germany, 40225, Düsseldorf, North Rhine-Westphalia, Germany